CLINICAL TRIAL: NCT01054183
Title: The Use of the GlideScope Ranger in Pediatric Critical Care Transport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090903
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Respiratory Failure
Keywords: respiratory failure, intubation, GlideScope, pediatric
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation using GlideScope Ranger (Experimental): The study site has two critical care transport teams per shift and will, at shift change, assign intubation team A to use the GlideScope Ranger for all intubations on that day.
  Interventions: Device: GlideScope Ranger Intubation
- intubation using direct laryngoscopy (Active Comparator): The study site has two critical care transport teams per shift and will, at shift change, assign intubation team B. Team B will do intubations using direct laryngoscopy only that day.
  Interventions: Device: Direct Laryngoscopy

INTERVENTIONS:
Device: GlideScope Ranger Intubation — Intubation with GlideScope Ranger Video Laryngoscope
  Arms: Intubation using GlideScope Ranger
Device: Direct Laryngoscopy — Intubations will be done with direct laryngoscopy.
  Arms: intubation using direct laryngoscopy

SUMMARY:
This study seeks to assess the role of the GlideScope Ranger video laryngoscope in facilitating successful neonatal/pediatric intubation by pediatric critical care transport teams. The central hypothesis of this study is that the GlideScope Ranger video laryngoscope reduces the rates of failed intubation attempts by pediatric critical care transport teams. The aims of this project are designed to specifically: (1) Establish competencies for GlideScope Ranger video laryngoscopy-assisted intubation for pediatric and neonatal patients; and (2) Compare the intubation success rates for intubation using GlideScope Ranger video laryngoscopy and using conventional, direct laryngoscopy by pediatric and neonatal critical care transport teams.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years
* Presence of respiratory failure requiring tracheal intubation by the Critical Care Transport Team either at the referring institution or during the transport to the receiving institution
* Ability of parent or legal guardian to provide written informed consent

Exclusion Criteria:

* Patients 18+ years of age
* Patient has a functioning tracheostomy
* Patient does not require orotracheal intubation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Bigham, M.D., Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Cooper RM. The GlideScope videolaryngoscope. Anaesthesia. 2005 Oct;60(10):1042. doi: 10.1111/j.1365-2044.2005.04384.x. No abstract available. PMID 16179054
- [Background] Lim TJ, Lim Y, Liu EH. Evaluation of ease of intubation with the GlideScope or Macintosh laryngoscope by anaesthetists in simulated easy and difficult laryngoscopy. Anaesthesia. 2005 Feb;60(2):180-3. doi: 10.1111/j.1365-2044.2004.04038.x. PMID 15644017
- [Background] Malik MA, O'Donoghue C, Carney J, Maharaj CH, Harte BH, Laffey JG. Comparison of the Glidescope, the Pentax AWS, and the Truview EVO2 with the Macintosh laryngoscope in experienced anaesthetists: a manikin study. Br J Anaesth. 2009 Jan;102(1):128-34. doi: 10.1093/bja/aen342. PMID 19059923
- [Background] Rai MR, Dering A, Verghese C. The Glidescope system: a clinical assessment of performance. Anaesthesia. 2005 Jan;60(1):60-4. doi: 10.1111/j.1365-2044.2004.04013.x. PMID 15601274
- [Background] Kim JT, Na HS, Bae JY, Kim DW, Kim HS, Kim CS, Kim SD. GlideScope video laryngoscope: a randomized clinical trial in 203 paediatric patients. Br J Anaesth. 2008 Oct;101(4):531-4. doi: 10.1093/bja/aen234. Epub 2008 Aug 8. PMID 18689807
- [Background] Milne AD, Dower AM, Hackmann T. Airway management using the pediatric GlideScope in a child with Goldenhar syndrome and atypical plasma cholinesterase. Paediatr Anaesth. 2007 May;17(5):484-7. doi: 10.1111/j.1460-9592.2006.02149.x. PMID 17474957
- [Background] Taub PJ, Silver L, Gooden CK. Use of the GlideScope for airway management in patients with craniofacial anomalies. Plast Reconstr Surg. 2008 Apr;121(4):237e-238e. doi: 10.1097/01.prs.0000305397.19883.a7. No abstract available. PMID 18349622
- [Background] Trevisanuto D, Fornaro E, Verghese C. The GlideScope video laryngoscope: initial experience in five neonates. Can J Anaesth. 2006 Apr;53(4):423-4. doi: 10.1007/BF03022520. No abstract available. PMID 16575049
- [Background] Nichols, D.G. and M.C. Rogers, Rogers' textbook of pediatric intensive care. 4th ed. 2008, Philadelpia: Lippincott Williams & Wilkins. No PMID Available.
- [Background] 04/14/2009 [cited 2009 June]; Available from: http://www.aap.org/sections/transmed/DatabaseTM.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospectively enrolled 22 patients between 8/1/2010 - 5/1/2012.
Pre-assignment Details: Prior to the initiation of the study, staff received didactic and simulation based instruction with the Glidescope Video Laryngoscope (GVL) and demonstrated competency through a minimum of 5 successful intubations in patients >10 kg and 1 intubation in a patient < or = 10 Kg in a controlled operating room setting.
Groups:
- GlideScope Ranger Intubation: The study site has two critical care transport teams per shift and will, at shift change, assign intubation team A to use the GlideScope Ranger for all intubations on that day.
  GlideScope Ranger Intubation : Intubation with GlideScope Ranger Video Laryngoscope
- Direct Laryngoscopy Intubation: The study site has two critical care transport teams per shift and will, at shift change, assign intubation team B. Team B will do intubations using direct laryngoscopy only that day.
  Direct Laryngoscopy : Intubations will be done with direct laryngoscopy.
Period: Overall Study
Arm/Group | GlideScope Ranger Intubation | Direct Laryngoscopy Intubation
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GlideScope Ranger Intubation | Direct Laryngoscopy Intubation | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.1 (4.56) | 1.5 (3.02) | 1.8 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Successful 1st Intubation Attempt
Description: Percent of participants with successful 1st intubation attempt by group (GVL vs. DL)
Time Frame: 30 days
Measure: Number; unit: Percent of Participants
Arm/Group | GlideScope Ranger Intubation | Direct Laryngoscopy Intubation
Number analyzed (Participants) | 10 | 12
Percent of Participants | 30 | 41.67
Statistical Analysis 1: Comparison: GlideScope Ranger Intubation vs Direct Laryngoscopy Intubation; Null hypothesis: the proportion of successful 1st intubation attempt is the same for both groups; Test type: Non-Inferiority or Equivalence — powered for 62 patients; p = 0.57, z test, two-sided

2. Primary Outcome: Overall Successful Intubation Rate: GlideScope Video Laryngoscopy (GVL) vs. Direct Laryngoscopy (DL).
Description: Overall successful intubation rate defined as all successful intubations (by type) divided by all attempts (by type).
Time Frame: 30 days; no long-term outcome measures were included
Population: The study was powered for 62 patients per study arm. Due to slow patient enrollment, the study was stopped prior to full enrollment with the aforementioned 22 total patients.
Measure: Number; unit: Percent of successful intubations
Units Other Than Participants: total intubation attempts
Arm/Group | GlideScope Ranger Intubation | Direct Laryngoscopy Intubation
Number analyzed (Participants) | 10 | 12
Number analyzed (total intubation attempts) | 19 | 28
Percent of successful intubations | 26.3 | 64.3
Statistical Analysis 1: Comparison: GlideScope Ranger Intubation vs Direct Laryngoscopy Intubation; Null hypothesis: overall successful intubation rate is the same for both groups; Test type: Non-Inferiority or Equivalence — powered for 62 patients; p = 0.002, z test, two-sided

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- GlideScope Video Laryngoscope Ranger(GVL): Procedure used to perform tracheal intubation that facilitates indirect visualization of the glottis through a video display.
- Direct Laryngoscopy: Procedure used to visualize the vocal cords and perform tracheal intubation in the pediatric and neonatal population.
Arm/Group | GlideScope Video Laryngoscope Ranger(GVL) | Direct Laryngoscopy
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 6/10 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GlideScope Video Laryngoscope Ranger(GVL) (N=10) | Direct Laryngoscopy (N=12)
Secretions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Insufficient view (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Difficult passing ETT with stylet (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Patient movement (Nervous system disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Wrong size blade (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tube size inappropriate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The biggest limitation was slow patient enrollment, prompting the study to be closed prior to reaching the full study power. All data were reliably reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes